CLINICAL TRIAL: NCT05197972
Title: Phase III Study Evaluating a Non-drug Intervention (NDI) Program by Fixed-frequency Guided Breathing (Cardiac Coherence) Associated With Medical Hypnosis on Preoperative Anxiety in Oncological Surgery
Brief Title: Assessment of Cardiac Coherence Associated With Medical Hypnosis on Preoperative Anxiety in Oncological Surgery
Acronym: COHEC2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2021-09 COH; 2021-A01524-37 (Registry Identifier: ID RCB)
Record Dates: First submitted 2021-12-08; First posted 2022-01-20 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Surgery; Oncology
MeSH Terms: conditions — Neoplasms | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Control group : classic management of the preoperative period Experimental group: classic management of the preoperative period with a cardiac coherence program coupled with hypnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Classic management of the preoperative period with a cardiac coherence program coupled with hypnosis.
  Interventions: Other: cardiac coherence program coupled with hypnosis
- Control group (No Intervention): Classic management of the preoperative period

INTERVENTIONS:
Other: cardiac coherence program coupled with hypnosis — At home the patient will perform the cardiac coherence sessions between 7 days and a maximum of 15 days before the surgery through the application "Respirelax": 3 sessions per day, lasting 5 minutes with a breathing frequency of 6 cycles/min for a period of 7 days minimum and maximum 15 days.
  An audio tape read in a hypnotic tone can be listened to by the patient during the cardiac coherence program or at another time of the day (see the text of the audio tape).
  Arms: Experimental group

SUMMARY:
The investigator proposes to use the cardiac coherence technique (Cardiac Coherence) coupled with a hypnosis session to reduce pre-operative anxiety.

DETAILED DESCRIPTION:
The perioperative period is recognized as anxiety-provoking for most patients. In oncology, 60 to 80% of patients suffer from stress throughout their treatment. If for some patients, this anxiety is more or less manageable, for others, it is the major concern with regard to their intervention.

For many years, pharmacological premedication, especially with benzodiazepines, has been the gold standard for the treatment of preoperative anxiety, but this systematic prescription is increasingly controversial, especially in populations most exposed to side effects, such as elderly subjects and patients with cardiac or respiratory pathologies.

The aim of this study is to propose an alternative to pharmacological premedication by a non-drug approach.

The two techniques (the Fixed Rate Guided Breathing Technique = cardiac coherence and hypnosis) can potentiate each other and become synergistic. Thus, for patients undergoing oncological surgery, regular practice of cardiac coherence coupled with hypnosis prior to their surgery should enable them to better manage perioperative anxiety and thus significantly reduce their level of anxiety on the day of their surgery.

The association of the 2 techniques combines several advantages:

* It is totally "physiological", free and immediately available for the patient and without any undesirable effect;
* It gives autonomy to the patient to manage his stress, making him independent of chemical molecules, the presence of a third party or expensive equipment.
* It will allow oncology patients to use it throughout their care (invasive examinations, MRI imaging, heavy and complex care such as certain dressings, etc.)

This work will allow:

* To give oncology patients the possibility to be actors of their care by a self-management of their anxiety in substitution or complement of a medicated approach;
* To map anxiety in oncology surgery using a simple scale such as the EVA, which has not yet been done;
* To identify the most anxious patients in order to provide them with the appropriate management (pharmacological and/or NMI) before their surgery;
* To evaluate the correlation between the level of preoperative anxiety and the occurrence of postoperative adverse events;
* To evaluate the correlation between the level of anxiety and the quality of recovery (QoR) and the postoperative experience (EVAN-G).

Patients in the experimental group will be interviewed to explain how to perform the cardiac coherence and hypnosis sessions at home before the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patient with a scheduled surgery for a cancer (suspected or declared) with a classic or ambulatory hospitalization
3. Patients requiring general anesthesia with or without associated loco-regional anesthesia or loco-regional anesthesia alone
4. Patient with a smartphone or a tablet or a computer and able to install the application
5. Inclusion of the patient minimum 7 days before the date of the surgery
6. Patient who signed the informed consent
7. Patient affiliated to a French social security system

Exclusion Criteria:

1. Emergency surgery
2. Plastic surgery for reconstruction: lipomodelling
3. Prophylactic surgery: no suspected or existing cancer
4. Bradycardia (< 50 beats/minute) with β-blockers
5. Severe heart failure with ventricular ejection fraction < 40%
6. Uncontrolled chronic pain for more than three months on morphine
7. Patient with unstable epilepsy or respiratory pathology with rest dyspnea
8. Patient used to and having a regular and habitual practice of relaxation techniques such as yoga, hypnosis, sophrology, meditation, music therapy, virtual reality, ...
9. Medical (neurological, psychiatric, etc.) or psychological conditions not allow for participation in the protocol (completion of questionnaires and booklet, compliance with the cardiac coherence program coupled with hypnosis)
10. Deaf patient without hearing aids
11. Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) of global anxiety | The morning of the surgery (Day 0) upon arrival in the operating room
  Visual Analogue Scale (VAS) of global anxiety is a anxiety self-assessment scale that allows the patient to self-assess his or her anxiety using a cursor. The scale ranges from 0 (no anxiety) to 100 (maximum anxiety).

SECONDARY OUTCOMES:
Program compliance | Between -15 to -7 days before surgery (Day -15 to Day -7) until the day of surgery (Day 0)
  Program compliance rate of patients in the experimental group. A patient is considered compliant if he declares to have completed at least 2/3 of the proposed Cardiac Coherence sessions + listening to hypnotic tape (at least 5 days /7).
Measurement of global and specific anxiety level by using a Visual Analogue Scale (VAS) | Between -15 to -7 days before surgery (Day -15 to Day -7)
  Visual Analogue Scale (VAS) of anxiety is a anxiety self-assessment scale that allows the patient to self-assess his or her anxiety using a cursor. The scale ranges from 0 (no anxiety) to 100 (maximum anxiety). The patient assesses his global and specific anxiety related to: surgery, anesthesia, COVID infectious risk, fear of the unknown, oncological disease
Measurement of global anxiety level by using a Visual Analogue Scale (VAS) | Between -15 to -7 days before surgery and the day of surgery (Day 0)
  Visual Analogue Scale (VAS) of global anxiety is a anxiety self-assessment scale that allows the patient to self-assess his or her anxiety using a cursor. The scale ranges from 0 (no anxiety) to 100 (maximum anxiety).
The preoperative anxiety score by using the Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Between -15 to -7 days before surgery
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a self-report questionnaire comprising six questions that have been developed and validated to evaluate the preoperative anxiety of patients. This global index assesses three separate areas: anxiety about anaesthesia, anxiety about surgery, and the desire for information.
  The scale scores six items from 1 to 5 (1 = absence, 5 = extreme). The APAIS scale will be used to determine the psychological profile of patients between "blunting" and "monitoring" types
VAS values and individual psycho-clinical characteristics | Between -15 to -7 days before surgery and the day of surgery (Day 0)
  Visual Analogue Scale (VAS) of global anxiety is a anxiety self-assessment scale that allows the patient to self-assess his or her anxiety using a cursor. The scale ranges from 0 (no anxiety) to 100 (maximum anxiety) (defined as VAS at Day 0 ≥ 40), and individual psycho-clinical characteristics (gender, smoking, psychological questionnaires).
Number of patients taking benzodiazepine | The day after surgery (Day 1)
  Rate of patients taking benzodiazepines in the 2 groups
Number of days of hospitalization | The day after surgery (Day -1) and up to 1 month
  Length of hospital stay in the 2 groups
VAS values and mode of hospitalization and importance of the surgical procedure | The morning of the surgery (Day 0) upon arrival in the operating room
  Visual Analogue Scale (VAS) of global anxiety is a anxiety self-assessment scale that allows the patient to self-assess his or her anxiety using a cursor, and the mode of hospitalization (ambulatory or conventional) and the importance of the surgical procedure (minor, intermediate or major)
Doses of hypnotic and morphine drugs | During anesthetic induction (Day 0)
  Doses of hypnotic and morphine drugs administered during anesthetic induction (Day 0) in the 2 groups
Value of preoperative VAS and adverse events | The morning of the surgery (Day 0) upon arrival in the operating room
  Visual Analogue Scale (VAS) of global anxiety is a anxiety self-assessment scale that allows the patient to self-assess his or her anxiety using a cursor and adverse event variables: pain, agitation, postoperative nausea and vomiting (PONV), ...
Number of Self-questionnaire completed | From the day of the anesthesia consultation until the end of the study
  Self-questionnaire completion rates for each of the 2 pre- and postoperative periods
Evaluation of the Vecu of General Anesthesia questionnaire (EVAN-G) | Two day after surgery (Day 2)
  The EVAN-G questionnaire includes 26 questions whose results are grouped together to define 6 dimensions: Attention Focus, Information, Privacy, Pain, Discomfort and Wait Times. From these scores, an overall satisfaction score is calculated. The total score of the six dimensions reduced to 100.
Visual Analogue Scale (VAS) of pain | At 1, 2 and 3 month after surgery
  Visual Analogue Scale (VAS) of pain is a pain self-assessment scale that allows the patient to self-assess his or her pain using a cursor
Quality of Recovery (QoR) | The day after surgery (Day 1)
  The QoR-15 questionnaire assesses five dimensions of recovery : physical comfort; emotional state; physical independence; physiological support; and pain. Each item was rated on a ten-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score of 15 ranges from 0 (poorest quality of recovery) to 150 (best quality of recovery).
Insomnia Severity Index Scale (ISI) | The day after surgery (Day 1)
  The Insomnia Severity Index (ISI) includes 7 questions which assesses the nature of the insomnia, the person's satisfaction with sleep, daily functioning and anxiety about sleep problems. Add scores for all seven items, sum from 0-7 = No clinically significant insomnia to 22-28 = Clinical insomnia (severe).
VAS of on satisfaction with overall management and anesthesia | The day after surgery (Day 1)
  Visual Analogue Scale (VAS) of on satisfaction with overall management and anesthesia is a satisfaction self-assessment scale that allows the patient to self-assess his or her satisfaction using a cursor. The scale ranges from 0 (not at all satisfied) to 100 (completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jibba AMRAOUI, MD, Study Chair — Institut régional du cancer de Montpellier; Régis FUZIER, MD, Principal Investigator — Institut Universitaire du Cancer Toulouse - Oncopole; Lauriane Bordevane, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (4):
- France (4):
  - Institut régional du cancer de Montpellier, Montpellier, Hérault
  - Centre Léon Bérard, Lyon
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all de-identified participants' data, the study protocol, the statistical analysis plan and the clinical study report. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to study data upon written detailed request sent to ICM, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Pekcan M, Celebioglu B, Demir B, Saricaoglu F, Hascelik G, Yukselen MA, Basgul E, Aypar U. The effect of premedication on preoperative anxiety. Middle East J Anaesthesiol. 2005 Jun;18(2):421-33. PMID 16438017
- [Background] Shevde K, Panagopoulos G. A survey of 800 patients' knowledge, attitudes, and concerns regarding anesthesia. Anesth Analg. 1991 Aug;73(2):190-8. doi: 10.1213/00000539-199108000-00013. PMID 1854034
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Bandeira D, Ferreira MB. Risk factors for preoperative anxiety in adults. Acta Anaesthesiol Scand. 2001 Mar;45(3):298-307. doi: 10.1034/j.1399-6576.2001.045003298.x. PMID 11207465
- [Background] Miller SM. Coping with impending stress: psychophysiological and cognitive correlates of choice. Psychophysiology. 1979 Nov;16(6):572-81. doi: 10.1111/j.1469-8986.1979.tb01523.x. No abstract available. PMID 515298
- [Background] Miller SM, Mangan CE. Interacting effects of information and coping style in adapting to gynecologic stress: should the doctor tell all? J Pers Soc Psychol. 1983 Jul;45(1):223-36. doi: 10.1037//0022-3514.45.1.223. PMID 6886967
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Background] Jamison RN, Taft K, O'Hara JP, Ferrante FM. Psychosocial and pharmacologic predictors of satisfaction with intravenous patient-controlled analgesia. Anesth Analg. 1993 Jul;77(1):121-5. PMID 8317718
- [Background] Kulik JA, Mahler HI, Moore PJ. Social comparison and affiliation under threat: effects on recovery from major surgery. J Pers Soc Psychol. 1996 Nov;71(5):967-79. doi: 10.1037//0022-3514.71.5.967. PMID 8939044
- [Background] Munoz HR, Dagnino JA, Rufs JA, Bugedo GJ. Benzodiazepine premedication causes hypoxemia during spinal anesthesia in geriatric patients. Reg Anesth. 1992 May-Jun;17(3):139-42. PMID 1606095
- [Background] Agelink MW, Majewski TB, Andrich J, Mueck-Weymann M. Short-term effects of intravenous benzodiazepines on autonomic neurocardiac regulation in humans: a comparison between midazolam, diazepam, and lorazepam. Crit Care Med. 2002 May;30(5):997-1006. doi: 10.1097/00003246-200205000-00008. PMID 12006794
- [Background] Maurice-Szamburski A, Auquier P, Viarre-Oreal V, Cuvillon P, Carles M, Ripart J, Honore S, Triglia T, Loundou A, Leone M, Bruder N; PremedX Study Investigators. Effect of sedative premedication on patient experience after general anesthesia: a randomized clinical trial. JAMA. 2015 Mar 3;313(9):916-25. doi: 10.1001/jama.2015.1108. PMID 25734733
- [Background] Lehrer PM, Gevirtz R. Heart rate variability biofeedback: how and why does it work? Front Psychol. 2014 Jul 21;5:756. doi: 10.3389/fpsyg.2014.00756. eCollection 2014. PMID 25101026
- [Background] Jiang H, White MP, Greicius MD, Waelde LC, Spiegel D. Brain Activity and Functional Connectivity Associated with Hypnosis. Cereb Cortex. 2017 Aug 1;27(8):4083-4093. doi: 10.1093/cercor/bhw220. PMID 27469596
- [Background] McCraty R, Atkinson M, Tiller WA, Rein G, Watkins AD. The effects of emotions on short-term power spectrum analysis of heart rate variability. Am J Cardiol. 1995 Nov 15;76(14):1089-93. doi: 10.1016/s0002-9149(99)80309-9. PMID 7484873
- [Background] Amraoui J, Pouliquen C, Fraisse J, Dubourdieu J, Rey Dit Guzer S, Leclerc G, de Forges H, Jarlier M, Gutowski M, Bleuse JP, Janiszewski C, Diaz J, Cuvillon P. Effects of a Hypnosis Session Before General Anesthesia on Postoperative Outcomes in Patients Who Underwent Minor Breast Cancer Surgery: The HYPNOSEIN Randomized Clinical Trial. JAMA Netw Open. 2018 Aug 3;1(4):e181164. doi: 10.1001/jamanetworkopen.2018.1164. PMID 30646110
- [Derived] Amraoui J, Bordenave L, Leclerc G, Salvignol G, Jarlier M, Fiess C, Philibert L, Fuzier R, Touraine C. Benefits of cardiac coherence combined with medical hypnosis on preoperative anxiety before cancer surgery: the COHEC II study trial protocol. BMJ Open. 2023 Dec 12;13(12):e072215. doi: 10.1136/bmjopen-2023-072215. PMID 38086587
- See also: 2. Amouroux R, Rousseau-Salvador C, Annequin D. L'anxiété préopératoire: manifestations cliniques, évaluation et prévention. Ann Méd-PsycholRevPsychiatr; 2010; 168:588-92 — https://hal.archives-ouvertes.fr/hal-00682246/document
- See also: Servant D, Lebeau JC, Mouster Y et al. Cardiac variability, a good indicator of emotion regulation. Journal of cognitive behavioral therapy 2008; 18: 45-8. — https://www.em-consulte.com/article/177897/resume/la-variabilite-cardiaque-un-bon-indicateur-de-la-r
- See also: Robert B. Measurement of preoperative anxiety by the visual analog scale. UE7: Professional thesis for the State Diploma of nurse anesthetist. CHU Poitiers — http://docplayer.fr/183897750-Mesure-de-l-anxiete-preoperatoire-par-l-echelle-visuelle-analogique.html